CLINICAL TRIAL: NCT02933385
Title: Activate Your Health Program : A Workplace Healthy Lifestyle Program
Brief Title: Active Your Health: A Workplace Healthy Lifestyle Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Marie-Ève Mathieu, Associate professor, Université de Montréal
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: University of Montreal
Record Dates: First submitted 2016-10-05; First posted 2016-10-14 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Lifestyle; Exercise; Nutrition
MeSH Terms: conditions — Motor Activity | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: 5 options are offered, however one option was not chosen by the companies so 4 will be analyzed in future studies
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Full lifestyle program (Experimental): Participants receive all the intervention tools that aimed to enhance lifestyle profile.
  Interventions: Behavioral: Health Risks assessement; Behavioral: Web-based health discussions; Behavioral: SOScuisine website; Behavioral: Health screening; Behavioral: Closing events; Behavioral: Coaching; Behavioral: Social Health platform; Behavioral: Accelerometer provided
- High lifestyle program (Experimental): Participants receive most of the intervention tools that aimed to enhance lifestyle profile.
  Interventions: Behavioral: Health Risks assessement; Behavioral: Web-based health discussions; Behavioral: SOScuisine website; Behavioral: Health screening; Behavioral: Closing events; Behavioral: Coaching; Behavioral: Social Health platform
- Moderate lifestyle program (Experimental): Participants receive some intervention tools that aimed to enhance lifestyle profile.
  Interventions: Behavioral: Health Risks assessement; Behavioral: Web-based health discussions; Behavioral: SOScuisine website; Behavioral: Closing events; Behavioral: Coaching
- Light lifestyle program (Experimental): Participants receive little intervention tools that aimed to enhance lifestyle profile.
  Interventions: Behavioral: Health Risks assessement; Behavioral: Web-based health discussions; Behavioral: SOScuisine website
- Control group (No Intervention): Participants receive none of the intervention tools that aimed to enhance lifestyle profile.

INTERVENTIONS:
Behavioral: Health Risks assessement — Home made questionnaire questioning about the participant's lifestyle habits, risk factors and other.
  Arms: Full lifestyle program; High lifestyle program; Light lifestyle program; Moderate lifestyle program
Behavioral: Web-based health discussions — Create interactions between the employees.
  Arms: Full lifestyle program; High lifestyle program; Light lifestyle program; Moderate lifestyle program
Behavioral: SOScuisine website — Site that is personalized to the employee. It provides menus, grocery shopping list and other.
  Arms: Full lifestyle program; High lifestyle program; Light lifestyle program; Moderate lifestyle program
Behavioral: Health screening — Screen for diabetes, cholesterol, blood pressure and body weight.
  Arms: Full lifestyle program; High lifestyle program
Behavioral: Closing events — these aim to motivate the employees to continue into the program.
  Arms: Full lifestyle program; High lifestyle program; Moderate lifestyle program
Behavioral: Coaching — The first year participant will be coached by a nurse, second year by a nutritionist, and third year by a kinesiologist.
  Arms: Full lifestyle program; High lifestyle program; Moderate lifestyle program
Behavioral: Social Health platform
  Arms: Full lifestyle program; High lifestyle program
Behavioral: Accelerometer provided — Social Health Platform: employees can challenge themselves or each other.
  Arms: Full lifestyle program

SUMMARY:
Currently there are very few studies that integrate classical interventions (screening clinics) and online tools in order to obtain sustainable lifestyle changes in workers efficiently. The current project aims to evaluate the efficiency of a combined approach versus the more traditional approach. Health Data collected by CAPSANA in the workplace between 2012 and 2014 showed that, out of 4231 workers, 69% should aim to do more active lifestyle and 74% to a better nutrition profile. In addition, 53% of the sampled population were overweight. In this context, the current project aims to motivate aims to motivate and follow individuals towards a healthier lifestyle. To do so, the Activate Your Health will be implemented and tested using various options (limited to more complete) in several companies.

DETAILED DESCRIPTION:
Currently, lifestyle habits of workers does not only represents a personal concern, but also a concern of the company. Currently there are very few studies that efficiently integrate classical interventions (screening) and online tools in order to obtain sustainable lifestyle changes in workers. The current project aims to evaluate efficacy of a combined approach versus more traditional approaches. Health Data collected by CAPSANA in the workplace between 2012 and 2014 showed that, out of 4231 workers, 69% should aim at a more active lifestyle and 74% at a better nutritional profile. In addition, 53% of the sampled population were overweight.

In this context, the current project aims to motivate and follow individuals towards a healthier lifestyle. To do so, the Activate Your Health will be implemented and tested using various options (limited to more complete) in several companies. It is planned to compare to a control group receiving no intervention to the other groups containing little to complete set of interventions. The content of the interventions involves health assessment, electronic tools (SOScuisine and social media platform), health screening, activity monitor tool and closing events. The companies had to pick which option they would like to provide their employees. It is anticipated that the complete option will yield better results for the activity profile and other lifestyle habits. For example, changes in eating habits toward better habits are expected.

ELIGIBILITY:
Inclusion Criteria:

* French Speaking, work in the participating company.

Exclusion Criteria:

* pregnant women.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2737 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity profile (intensity, frequency and duration) measured by questionnaire | 365 days
  Based on a questionnaire we will be able to calculate physical activity duration, intensity and frequency will be obtained.

SECONDARY OUTCOMES:
Nutritional profile (fruit and vegetables intake) will be obtained by questionnaire | 365 days
  Based on a questionnaire we will be able to calculate nutrition parameters (# of fruits and vegetables per day).

REFERENCES:
- [Derived] Kugathasan TA, Lecot F, Laberge S, Tremblay J, Mathieu ME. Activate Your Health, a 3-year, multi-site, workplace healthy lifestyle promotion program: study design. BMC Public Health. 2019 Aug 19;19(1):1140. doi: 10.1186/s12889-019-7393-x. PMID 31426771